CLINICAL TRIAL: NCT03618264
Title: Pre-emptive Scalp Infiltration With Dexamethasone Plus Ropivacaine vs. Ropivacaine for Relief of Postoperative Pain After Craniotomy in Adults
Brief Title: Pre-emptive Scalp Infiltration With Dexamethasone Plus Ropivacaine for Postoperative Pain After Craniotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY 2018-034-02-1
Record Dates: First submitted 2018-07-30; First posted 2018-08-07 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Pain, Postoperative; Post-Craniotomy Headache
Keywords: Postoperative Pain; Post-Craniotomy Headache; Dexamethasone; Ropivacaine; Pre-emptive Scalp Infiltration
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone plus Ropivacaine group (Experimental): Participates received peri-incisional scalp infiltration of a miscible liquid of dexamethasone and ropivacaine. The local infiltration miscible liquid containing 0.33mg dexamethasone and 5mg ropivacaine per milliliter
  Interventions: Drug: Miscible liquid of dexamethasone and ropivacaine
- Ropivacaine group (Active Comparator): Participates received peri-incisional scalp infiltration of 5mg/mL ropivacaine.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Miscible liquid of dexamethasone and ropivacaine — Intervention in this study will be peri-incisional scalp infiltration with dexamethasone, ropivacaine and normal saline miscible liquids for participants who will undergo elective craniotomy. The local infiltration solution containing 0.33mg dexamethasone and 5mg ropivacaine per milliliter will be infiltrated along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigator.
  Arms: Dexamethasone plus Ropivacaine group
Drug: Ropivacaine — Intervention in this study will be peri-incisional scalp infiltration with ropivacaine for participants who will undergo elective craniotomy. The local infiltration solution containing 5mg ropivacaine per milliliter will be infiltrated along the incision and throughout the entire thickness of the scalp before skin incision. The volume of local infiltration solution will be decided by surgeons according to the cut length, and the capacity of the solution will be recorded by investigator.
  Arms: Ropivacaine group

SUMMARY:
A majority of patients would suffer from moderate-to-severe postoperative pain after undergoing craniotomy. As a result, adequate pain control is essential for patients' prognosis and their postoperative life quality. Although opioids administration is regarded as the first-line analgesic for post-craniotomy pain management, it may be associated with delayed awakening, respiratory depression, hypercarbia and it may interfere with the neurologic examination. For the avoidance of side-effects of systemic opioids, local anesthetics administered around the incision have been performed clinically. However, some studies revealed that the analgesic effect of local anesthetics was not unsatisfactory due to its short pain relief duration. As is reported that postoperative pain of craniotomy is mainly caused by skin incision and reflection of muscles, preventing the liberation of inflammatory mediators around the incision seems to be more effective than simply blocking nerve conduction. Thus, Investigators suppose that pre-emptive scalp infiltration with steroid (dexamethasone) plus local anesthetic (ropivacaine) could relieve postoperative pain after craniotomy in adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective craniotomy for resection of a supratentorial tumour under general anaesthesia;
* American Society of Anesthesiologists (ASA) physical status of I or II;
* Participates required to fix their head in a head clamp intraoperatively;
* Participates with an anticipated fully recovery within 2 hours postoperatively.

Exclusion Criteria:

* History of craniotomy;
* Expected delayed extubation or no plan to extubate;
* Participants who cannot use a patient-controlled analgesia (PCA) device;
* Participants who cannot understand the instructions of a numeral rating scale (NRS) 35 before surgery;
* Extreme body mass index (BMI) (< 15 or > 35);
* Allergy to opioids, dexamethasone or ropivacaine;
* History of excessive alcohol or drug abuse, chronic opioid use (more than 2 weeks), or use of drugs with confirmed or suspected sedative or analgesic effects;
* History of psychiatric disorders, uncontrolled epilepsy or chronic headache;
* Pregnant or at breastfeeding;
* Symptomatic cardiopulmonary, renal, or liver dysfunction or history of diabetes;
* Preoperative Glasgow Coma Scale< 15;
* Suspicion of intracranial hypertension;
* Peri-incisional infection;
* Participants who have received radiation therapy and chemotherapy preoperatively or with a high probability to require a postoperative radiation therapy and chemotherapy according to the preoperative imaging.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Cumulative sufentanil consumption within 48 hours postoperatively | Within 48 hours after the operation
  All participates will receive an electronic intravenous patient-controlled analgesia (PCA) device in which the bolus dose of sufentanil will be set as 2 μg with a lockout interval of 10 min and the maximum dose will be limited as 8 μg per hour. If the participates feel inadequate analgesia after 5 times of sufentanil bolus, the bolus dose will be increased to 3 μg and the maximum dose will be increased to 12 μg per hour.

SECONDARY OUTCOMES:
The number of participants who have no sufentanil consumption | Within 48 hours after the operation
  The number of participants who have not pushed the button of patient-controlled analgesia pump. Both of the initial dose and background infusion of the patient-controlled analgesia pump in this study will be set as 0. Participates will be advised to push the analgesic demand button if they feel pain.
The first time to press the patient-controlled analgesia button | Within 48 hours after the operation
  The first time that the participants press the patient-controlled analgesia button.
The total times that participants press patient-controlled analgesia button | Within 48 hours after the operation
  The total times that participants press patient-controlled analgesia button including effective presses and ineffective presses.
Numerical rating scale of pain | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks, 1 month, 3 months and 6 months after surgery
  Pain was assessed after surgery by a numerical rating scale (0 indicates no pain, 10 indicates the most severe pain imaginable).
Postoperative nausea and vomiting | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  Postoperative nausea and vomiting (PONV) was rated by participates as: 0, absent; 1, nausea not requiring treatment; 2, nausea requiring treatment; and 3, vomiting.
Ramsay Sedation Scale | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  Ramsey 1: Anxious, agitated, restless; Ramsey 2: Cooperative, oriented, tranquil; Ramsey 3: Responsive to commands only If Asleep; Ramsey 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsey 5: Sluggish response to light glabellar tap or loud auditory stimulus; Ramsey 6: No response to light glabellar tap or loud auditory stimulus
Respiratory depression | Within 48 hours after the operation
  Respiratory depression is defined as a respiratory rate less than 10 breaths per minute or oxygen saturation was less than ninety percent.
Heart rate | Before anesthesia induction, after anesthesia induction, after scalp infiltration, during skull drilling, mater cutting, skin closure and at 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
Mean arterial pressure | Before anesthesia induction, after anesthesia induction, after scalp infiltration, during skull drilling, mater cutting, skin closure and at 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
The times of emergency reducing blood pressure after the operation | Within 48 hours after the operation
  The criteria for treatment is determined by the participant's surgeon in charge.The times of emergency reducing blood pressure will be recording by the investigator.
Patient satisfactory scale (PSS) | At 48 hours, 1 week, 1 month, 3 months and 6 months after surgery
  0 for unsatisfactory, and 10 for very satisfied
The total consumption of opioids during the operation | During procedure
The total consumption of anaesthetic during the operation | During procedure
The duration of hospitalization after the operation | Approximately 2 weeks after the operation
The World Health Organization Quality of Life (WHOQOL)-BREF | At 1 month, 3 months and 6 months after surgery
  Quality of life will be measured using the World Health Organisation QoL-BREF (WHOQOL-BREF) questionnaire. The WHOQOL-BREF is a abbreviated version of the WHOQOL-100 assessment. WHOQOL-BREF is a self-report questionnaire that contains 26 items and addresses 4 QOL domains: physical health (7 items), psychological health (6 items), social relationships (3 items) and environment (8 items). Two other items measure overall QOL and general health. Each domain's mean score can range between 4 and 20 and a higher score indicates a higher quality of life. The mean score of items within each domain is used to calculate the domain score. A transformation method converts domain scores to a 0-100 scale.
Incisional related adverse events Incisional related adverse events | Within 1 month after surgery
  Including delayed incisional healing, incisional infection, intracranial infection, scar healing
Wound Healing Score | At 3 weeks and 6 weeks after surgery
  Skin Healing
  1: fully healed; 2: ≤3 cm in total not healed; 3: >3 cm not healed; 4: areas of necrosis ≤3 cm; 5: areas of necrosis >3 cm Infection
  1: none; 2: ≤0.5-cm margin of redness; 3: more redness or superficial pus; 4: deep infection; not applicable Hair Regrowth
  1: even regrowth along wound; 2: ≤3 cm not regrowing; 3: >3-6 cm not regrowing; 4: >6 cm not regrowing; not applicable
Patient and Observer Scar Assessment Scale | At 6 months after surgery
  The Patient and Observer Scar Assessment Scale includes subjective symptoms of pain and pruritus and consists of 2 numerical numeric scales: The Patient Scar Assessment Scale and the Observer Scar Assessment Scale. It assesses vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion for a scar on a score of 1 (normal skin) to 10 (worst scar imaginable). and it incorporates patient assessments of pain, itching, color, stiffness, thickness, relief and overall opinion. Participants were asked to rate the severity of their scar compared to normal skin. The overall opinion scale score ranged from 1 (normal skin) to 10 (very different from normal skin).

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rocha-Filho PA. Post-craniotomy headache: a clinical view with a focus on the persistent form. Headache. 2015 May;55(5):733-8. doi: 10.1111/head.12563. Epub 2015 Apr 22. PMID 25903913
- [Background] Vallapu S, Panda NB, Samagh N, Bharti N. Efficacy of Dexmedetomidine as an Adjuvant to Local Anesthetic Agent in Scalp Block and Scalp Infiltration to Control Postcraniotomy Pain: A Double-Blind Randomized Trial. J Neurosci Rural Pract. 2018 Jan-Mar;9(1):73-79. doi: 10.4103/jnrp.jnrp_310_17. PMID 29456348
- [Background] Tsaousi GG, Logan SW, Bilotta F. Postoperative Pain Control Following Craniotomy: A Systematic Review of Recent Clinical Literature. Pain Pract. 2017 Sep;17(7):968-981. doi: 10.1111/papr.12548. Epub 2017 Feb 23. PMID 27996204
- [Background] Chowdhury T, Garg R, Sheshadri V, Venkatraghavan L, Bergese SD, Cappellani RB, Schaller B. Perioperative Factors Contributing the Post-Craniotomy Pain: A Synthesis of Concepts. Front Med (Lausanne). 2017 Mar 1;4:23. doi: 10.3389/fmed.2017.00023. eCollection 2017. PMID 28299313
- [Background] Akcil EF, Dilmen OK, Vehid H, Ibisoglu LS, Tunali Y. Which one is more effective for analgesia in infratentorial craniotomy? The scalp block or local anesthetic infiltration. Clin Neurol Neurosurg. 2017 Mar;154:98-103. doi: 10.1016/j.clineuro.2017.01.018. Epub 2017 Jan 30. PMID 28183036
- [Background] Dunn LK, Naik BI, Nemergut EC, Durieux ME. Post-Craniotomy Pain Management: Beyond Opioids. Curr Neurol Neurosci Rep. 2016 Oct;16(10):93. doi: 10.1007/s11910-016-0693-y. PMID 27604271
- [Background] Mordhorst C, Latz B, Kerz T, Wisser G, Schmidt A, Schneider A, Jahn-Eimermacher A, Werner C, Engelhard K. Prospective assessment of postoperative pain after craniotomy. J Neurosurg Anesthesiol. 2010 Jul;22(3):202-6. doi: 10.1097/ANA.0b013e3181df0600. PMID 20479664
- [Background] Rahimi SY, Alleyne CH, Vernier E, Witcher MR, Vender JR. Postoperative pain management with tramadol after craniotomy: evaluation and cost analysis. J Neurosurg. 2010 Feb;112(2):268-72. doi: 10.3171/2008.9.17689. PMID 19630495
- [Background] Misra S, Koshy T, Suneel PR. Oral clonidine attenuates the fall in mean arterial pressure due to scalp infiltration with epinephrine-lidocaine solution in patients undergoing craniotomy: a prospective, randomized, double-blind, and placebo controlled trial. J Neurosurg Anesthesiol. 2009 Oct;21(4):297-301. doi: 10.1097/ANA.0b013e3181ac7a31. PMID 19955891
- [Derived] Zhao C, Wang S, Pan Y, Ji N, Luo F. Pre-Emptive Incision-Site Infiltration with Ropivacaine Plus Dexamethasone for Postoperative Pain After Supratentorial Craniotomy: A Prospective Randomized Controlled Trial. J Pain Res. 2021 Apr 19;14:1071-1082. doi: 10.2147/JPR.S300943. eCollection 2021. PMID 33907455